CLINICAL TRIAL: NCT02469415
Title: Phase II Study of Pacritinib for Patients With Lower-Risk Myelodysplastic Syndromes
Brief Title: Pacritinib for Patients With Lower-Risk Myelodysplastic Syndromes (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: FDA Clinical Hold
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: CTI BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0224; NCI-2015-01306 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-06-10; First posted 2015-06-11 (Estimated); Results first posted 2018-04-23 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-05

CONDITIONS: Leukemia
Keywords: Leukemia; Myelodysplastic syndromes; MDS; Lower-risk; Pacritinib; 5-azacitidine; Azacitidine; 5-azacytidine; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine; Decitabine; Dacogen
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Azacitidine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pacritinib + Azacitidine or Decitabine (Experimental): Part 1: Pacritinib 200 mg taken by mouth twice daily. Study cycles administered every 28 days.
  Part 2: After 4 cycles of treatment, Pacritinib combined with 5-azacitidine or Decitabine. Pacritinib decreased to 200 mg in morning and 100 mg in evening for first cycle of combined therapy with Pacritinib increased to 200 mg twice a day on subsequent cycles of combined therapy. Those with disease progression prior to 4 cycles of Pacritinib may initiate Pacritinib + HMA study portion prior to completion of 4 cycles. Starting dose of either 5-azacitidine 75 mg/m2 by vein (IV) or Decitabine 20 mg/m2 IVon Days 1 - 5 of Cycles 5 and beyond.
  Interventions: Drug: Pacritinib; Drug: 5-azacitidine; Drug: Decitabine

INTERVENTIONS:
Drug: Pacritinib — Part 1: Pacritinib 200 mg taken by mouth twice daily.
  Part 2: Pacritinib dose decreased to 200 mg in the morning and 100 mg in the evening for the first cycle of combined therapy. If no toxicity is observed in first cycle of combined therapy, Pacritinib dose may be increased to 200 mg twice a day on subsequent cycles of combined therapy.
Drug: 5-azacitidine — Part 2 Starting Dose of 5-azacitidine: 75 mg/m2 by vein on Days 1 - 5 of Cycles 5 and beyond.
  Other Names: Azacitidine; 5-azacytidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
Drug: Decitabine — Part 2 Starting Dose of Decitabine: 20 mg/m2 by vein on on Days 1 - 7 of Cycles 5 and beyond.
  Other Names: Dacogen

SUMMARY:
The goal of this clinical research study is to learn if pacritinib, either alone or in combination with azacitidine or decitabine, can help to control MDS.

The safety of this drug and drug combination will also be studied.

DETAILED DESCRIPTION:
Study Drug Administration:

Each cycle is 28 days.

If you are found to be eligible to take part in this study, you will take pacritinib by mouth 2 times each day during Cycles 1-4. Each dose should be about 12 hours apart (1 dose in the morning, 1 dose in the evening).

After Cycle 4, if the study doctor thinks it is in your best interest, you may be able to continue taking pacritinib in combination with either azacitidine or decitabine. The study doctor will tell you which drug you will receive. The study doctor will tell you which drug you will receive. Decitabine and azacitidine may be administered by local doctor or at MD Anderson. Cycle 1 of Part 2 will be administered at MD Anderson. Commercial supplies of decitabine and azacitidine will be used.

You will receive either azacitidine by vein over about 1 hour on Days 1-5 of Cycles 5 and beyond or decitabine by vein over about 1 hour or as an injection under the skin on Days 1-7 of Cycles 5 and beyond.

You should return any unused study drug and/or any empty bottles to each study visit.

Study Visits:

One (1) time each week during Cycle 1 and then on Day 1 of each cycle after that, blood (about 1½ teaspoons) will be drawn for routine tests. You may have this blood drawn at a local lab or clinic closer to your home, if the study doctor thinks this is acceptable. The results from the blood draw will be sent to the study doctor.

On Day 28 (+/- 5 days) of Cycles 1 and 4, you will have a bone marrow aspiration/biopsy to check for genetic mutations and cytogenetic testing. If you begin receiving pacritinib in combination with either azacitidine or decitabine, you will also have this test repeated at Cycle 4 of your combination therapy.

On Day 1 of Cycle 1, Day 28 of Cycles 1 and 4, and at any time the doctor thinks it is needed, you will have an EKG.

Length of Treatment:

You may continue taking pacritinib for up to 4 cycles. If the doctor thinks it is in your best interest, you may be eligible to continue taking the study drug in combination with either azacitidine or decitabine for as long as the doctor thinks it is in your best interest.

You will no longer be able to take the study drug(s) if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the end-of-treatment visit.

After the end of therapy and/or 30 days after your last dose of study drug, the study staff will follow your health status by phone call every 2 months (+/- 2 months) until you receive another cancer treatment.

End-of-Treatment Visit:

About 28 days after the last dose of study drug(s):

* Blood (about 1½ teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you will have a bone marrow aspirate/biopsy to check the status of the disease.

This is an investigational study. Pacritinib is not FDA approved or commercially available. It is currently being used for research purposes only. Azacitidine and decitabine are both FDA approved and commercially available for the treatment of MDS. The study doctor can explain how the study drugs are designed to work.

Up to 40 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent indicating that patients are aware of the investigational nature of this study, in keeping with the policies of MD Anderson Cancer Center (MDACC), must be obtained prior to any study specific procedures.
2. Patients with a histologically confirmed diagnosis of MDS by World Health Organization (WHO) classification, and lower-risk MDS as defined by the IPSS classification (Low or Int-1 disease) or R-IPSS classification (Very Low or Low) are eligible. Patients with MDS/MPD overlap syndromes including CMML are also eligible if they have Low or Int-1 disease per IPSS. Patients may have received MDS-directed therapy (i.e. lenalidomide), although patients with prior exposure to hypomethylating agents (e.g. 5-azacitidine or decitabine) are not eligible.
3. The interval from prior treatment to time of study drug administration is at least 1 week (except for hydroxyurea or steroid therapy) with recovery from all prior therapy-related toxicities
4. Age >/= 18 years old.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
6. Adequate liver function, as evidence by serum bilirubin </= 2x the laboratory normal range (except for patients with Gilbert's Disease) or an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) of </= 2.5x the upper limit of normal (ULN) or </= 5x ULN if hepatic disease involvement is present as determined by the investigator.
7. Serum creatinine (Cr) </= 2x ULN or 24-hour creatinine clearance >/=50 ml/min
8. Subjects of reproductive potential must agree to the use of acceptable contraceptive methods for the duration of the time on study and a further 6 months after completion of treatment. Women of childbearing potential must have a negative blood or urine pregnancy test within 72 hours of start of treatment.

Exclusion Criteria:

1. Subjects with any prior exposure to the hypomethylating agents (5-azacitidine or decitabine) are excluded.
2. Subjects with any prior exposure to JAK2 inhibitor therapy (i.e. ruxolitinib or prior pacritinib therapy) are excluded.
3. Any prior or coexisting medical condition that in the investigator's judgment will substantially increase the risk associated with the subject's participation in the study.
4. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures.
5. Active uncontrolled serious infection or sepsis at study enrollment. Patients receiving antibiotics for infections that are under control may be included in the study.
6. Gastrointestinal disorders that may significantly interfere with absorption of study drug.
7. Subjects have received potent CYP3A inhibitors within 7 days prior to the initiation of study treatment.
8. History of myocardial infarction, severe/unstable angina, or symptomatic congestive heart failure (New York Heart Failure (NYHA) Class III or IV congestive heart failure) within 6 months prior to study enrollment or Left ventricular ejection fraction (LVEF) <50%
9. Impaired cardiac function including ongoing cardiac dysrhythmias of Grade > 2, ejection fraction < 50%, atrial fibrillation of any grade, or QTc prolongation > 450 ms, or other factors that increase the risk of QT prolongation (i.e. family history of long QT interval syndrome, hypokalemia defined as serum potassium < 3.0 mEq/L)
10. Diagnosis of other malignancies within the last 3 years other than curatively treated non-melanoma skin cancer, carcinoma in situ of the cervix, organ-confined or treated non-metastatic prostate cancer, in situ breast carcinoma after complete surgical resection, or superficial transitional cell bladder carcinoma.
11. Known active Hepatitis A, B or C.
12. Known HIV seropositivity.
13. Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2017-06-03 (Actual); Study Completion 2017-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney DiNardo, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 2015 through February 2016. This study was closed by the FDA due to the Pacritinib hold. The study was closed to new patients February 10, 2016. All active patients were required to come off treatment at that time.
Pre-assignment Details: Three participants were registered on this study. One participant withdrew consent before receiving the study medication. Two participants were taken off study when the investigational agent was placed on full clinical hold by the Food and Drug Administration (FDA).
Groups:
- Pacritinib + Azacitidine or Decitabine: Pacritinib: Part 1: Pacritinib 200 mg taken by mouth twice daily.
  Part 2: Pacritinib dose decreased to 200 mg in the morning and 100 mg in the evening for the first cycle of combined therapy. If no toxicity is observed in first cycle of combined therapy, Pacritinib dose may be increased to 200 mg twice a day on subsequent cycles of combined t
Period: Overall Study
Arm/Group | Pacritinib + Azacitidine or Decitabine
Started | 3
Completed | 0
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Investigational agent placed on hold | 2

BASELINE CHARACTERISTICS:
Groups:
- Pacritinib + Azacitidine or Decitabine: Pacritinib: Part 1: Pacritinib 200 mg taken by mouth twice daily.
  Part 2: Pacritinib dose decreased to 200 mg in the morning and 100 mg in the evening for the first cycle of combined therapy. If no toxicity is observed in first cycle of combined therapy, Pacritinib dose may be increased to 200 mg twice a day on subsequent cycles of combined therapy.
  5-azacitidine: Part 2 Starting Dose of 5-azacitidine: 75 mg/m2 by vein on Days 1 - 5 of Cycles 5 and beyond.
  Decitabine: Part 2 Starting Dose of Decitabine: 20 mg/m2 by vein on on Days 1 - 7 of Cycles 5 and beyond.
Arm/Group | Pacritinib + Azacitidine or Decitabine
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 52 [52 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: The primary efficacy outcome of both parts is the overall response rate (ORR) based mainly on hematologic improvement defined by (International Working Group) IWG-2006 criteria, and which also includes complete remission (CR), partial remission (PR) and marrow complete remission.
Time Frame: 28 days
Population: Two participants were taken off study when the investigational agent was placed on full clinical hold by the Food and Drug Administration (FDA). The two participants who received the study medication were not on study long enough to make a formal response assessment.
Arm/Group | Pacritinib + Azacitidine or Decitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Participants will be assessed for adverse events from the first dose of study medication to the completion of study treatment, for up to 12 months.
Arm/Group | Pacritinib + Azacitidine or Decitabine
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pacritinib + Azacitidine or Decitabine (N=3)
Pneumonia (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-20): https://cdn.clinicaltrials.gov/large-docs/15/NCT02469415/Prot_SAP_000.pdf